CLINICAL TRIAL: NCT03847415
Title: Endometrial Evaluation in Cases of Postmenopausal Bleeding Using Three Dimensional Ultrasound , Power Doppler Angiography and Office Hysteroscopy in Correlation to Pathological Findings .
Brief Title: Endometrial Evaluation in Cases of Postmenopausal Bleeding
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed reda, assisant lecturer, Cairo University
Other Study IDs: endometrial volume
Record Dates: First submitted 2019-02-09; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Postmenopausal Bleeding
MeSH Terms: interventions — Ultrasonography; Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — to evalute abnormal uterine bleeding in postmenopausal women using 3D(dimensional) ultrasound assessment of endometrial volume .Doppler assessment of endometrium and hysteroscopy and to correlate this finding with pathological finding of endometrial biopsy
  Other Names: hysteroscopy; fractional currettage

SUMMARY:
The aim of this prospective observational study is to evaluate abnormal uterine bleeding in postmenopausal women using 3D(dimensional) ultrasound assessment of endometrial volume .Doppler assessment of endometrium and hysteroscopy and to correlate this finding with pathological finding of endometrial biopsy

DETAILED DESCRIPTION:
Postmenopausal bleeding (PMB) is defined as vaginal bleeding occurring after twelve months of amenorrhoea, in a woman of the age where the menopause can be expected. Hence it does not apply to a young woman, who has had amenorrhoea from anorexia nervosa, or a pregnancy followed by lactation. However, it can apply to younger women following premature ovarian failure or premature menopause, Postmenopausal bleeding is a common problem representing 5% of all gynaecology outpatient attendances. postmenopausal bleeding is usually the first symptom of endometrial cancer and active intervention can lead to its early detection. So, there is need of a diagnostic tool with high accuracy for detection of endometrial pathology in most efficient and least invasive method possible.

Endometrial sampling is the gold standard for diagnosing abnormalities in the endometrial tissues ,however . There is a growing trend to use noninvasive procedures such as TVS, to measure the endometrial thickness, diagnose adenomyosis, endometrial polyps .Another important ability of 3D TVS is volume calculation using the Virtual Organ Computer-aided AnaLysis (VOCAL) even in irregularly shaped structures. This method has been demonstrated to be more accurate than 2D-volume estimation .

• Hysteroscopy has the advantage of directly visualizing the uterine cavity and the endometrium, allowing biopsy to be taken immediately from the suspected abnormality.

ELIGIBILITY:
* Inclusion Criteria:
* Women Age > 45 years
* with postmenopausal uterine bleeding

Exclusion Criteria:

* Women with bleeding disorders or coagulopathy
* women with cervical cancer or breast carcinoma .
* history of tamoxifen intake
* women with fibroid .

Min Age: 45 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women Age > 45 years postmenopausal uterine bleeding
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
accuracy of 3d ultrasound in post menopausal bleeding | 6months
  to evalute women with postmenpausal uterine bleeding using three dimensional ultrasound assessment of endometrial volume

SECONDARY OUTCOMES:
comparison between hysteroscopy and ultrasound in post menopausal bleeding | 6months
  to compare hysteroscopy with ultrasound

REFERENCES:
- [Background] Goldstein SR. Modern evaluation of the endometrium. Obstet Gynecol. 2010 Jul;116(1):168-176. doi: 10.1097/AOG.0b013e3181dfd557. PMID 20567184
- [Background] Jacobs I, Gentry-Maharaj A, Burnell M, Manchanda R, Singh N, Sharma A, Ryan A, Seif MW, Amso NN, Turner G, Brunell C, Fletcher G, Rangar R, Ford K, Godfrey K, Lopes A, Oram D, Herod J, Williamson K, Scott I, Jenkins H, Mould T, Woolas R, Murdoch J, Dobbs S, Leeson S, Cruickshank D, Skates SJ, Fallowfield L, Parmar M, Campbell S, Menon U. Sensitivity of transvaginal ultrasound screening for endometrial cancer in postmenopausal women: a case-control study within the UKCTOCS cohort. Lancet Oncol. 2011 Jan;12(1):38-48. doi: 10.1016/S1470-2045(10)70268-0. Epub 2010 Dec 10. PMID 21147030